CLINICAL TRIAL: NCT00911638
Title: Are Patient Decision Aids for Total Joint Replacement Cost-effective and do They Optimize the Surgical Referral Process From Primary Care?
Brief Title: Comparison of Ways to Prepare Patients for Decisions About Joint Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other); The Ottawa Hospital (Other); Queensway Carleton Hospital (Other); University of Ottawa (Other); University of Toronto (Other); University of Chicago (Other); Northwestern University Feinberg School of Medicine (Other); Northwestern University (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OHRI-2006724; FIMDM Research Grant 0099-1 (Other Grant/Funding Number: FIMDM Research Grant 0099-1)
Record Dates: First submitted 2009-05-29; First posted 2009-06-02 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis
Keywords: Patient decision aids; Patient preferences; Osteoarthritis; Joint replacement; Waiting times
MeSH Terms: conditions — Osteoarthritis; Patient Preference

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Patient decision aid (Experimental): Patient decision aid focused on treatment options for osteoarthritis of the hip or knee and preference report for surgeons. The patient decision aid used is from the Informed Medical Decisions Foundation
  Interventions: Behavioral: Patient decision aid; Behavioral: Usual care
- 2: Usual care (Active Comparator): Usual patient educational resources for patients undergoing hip or knee replacement surgery.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Patient decision aid — Patients will receive i) Patient education:usual take home education brochure from recruiting hospital ii)a video/DVD PtDA for either hip (Treatment choices for hip osteoarthritis) or knee (Treatment choices for knee osteoarthritis) © Health Dialog 2005.
  iii) a personal decision form:an interactive form used by patients after the DVD to elicit their knowledge, values, preferred option, and perceptions of the decision making process.
  iv) Referred onward to the surgeon with their preferences for surgery using a standardized report of their clinical findings plus decisional data (knowledge, values, preference).
  Other Names: non applicable
  Arms: 1: Patient decision aid
Behavioral: Usual care — Patients will receive i) the usual take-home educational brochure available at the recruiting hospital describing preparation for surgery after the decision is made, recovery after surgery, and discharge plans.
  ii) Referral onward to surgeon with a standardized report of clinical findings only
  Other Names: non applicable

SUMMARY:
Ministries of Health consider wait lists for total joint replacement a top priority. Research priorities to manage wait lists indicate the need to establish benchmarks that consider patient preferences. However, patients' preferences for hip or knee replacements are strongly associated with their misperceptions of the indicators for, and the risks and benefits of, these procedures. These misperceptions can be corrected with the use of patient decision aids. When decision aids are used in combination with assessing surgical eligibility, there may be a reduction in unnecessary referrals for surgery either because the patient is ineligible or because the eligible candidates make informed decisions to forgo this option. The primary study objective is to evaluate the effect of patient decision aids (PtDAs) on total wait times (wait times for surgical consultation, plus wait times for surgery) when used in combination with a general practitioner run clinic to screen patients with hip or knee osteoarthritis for surgical eligibility. Major secondary objectives include determining (a) the effect of PtDAs on surgery rates within two years, (b) the effect of PtDAs on decision quality, and (c) cost-effectiveness of PtDAs for total joint arthroplasty.

DETAILED DESCRIPTION:
This was not indicated as required.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for surgical consultation for hip or knee osteoarthritis
* WOMAC and HKPT scores indicate that pain and functional criteria are rated as moderate or severe, or there is radiographic evidence of joint damage

Exclusion Criteria:

* Patients with inflammatory arthritis
* Patients who have had previous TJA
* Patients unable to understand video/DVD decision aids due to deafness, blindness, cognitive impairment, or language barrier

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2008-05; Primary Completion 2012-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Total wait time for surgery | September 2010

SECONDARY OUTCOMES:
Surgery rates determined by the proportion of patients who proceed to surgery within 2 years | January 2012
Decision quality, the extent to which patients decisions are informed and values-based | September 2010
Cost effectiveness (including estimated effects on quality adjusted life expectancy and costs) | December 2017
  This phase was delayed to have 5 years of follow-up data on all participants

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Stacey, RN PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - Queensway Carleton Hospital, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stacey D, Hawker G, Dervin G, Tomek I, Cochran N, Tugwell P, O'Connor AM. Management of Chronic Pain: Improving shared decision making in osteoarthritis. BMJ. 2008 Apr 26;336(7650):954-5. doi: 10.1136/bmj.39520.701748.94. Epub 2008 Apr 8. PMID 18397937
- [Background] Stacey D, Hawker G, Dervin G, Tugwell P, Boland L, Pomey MP, O'Connor AM, Taljaard M. Decision aid for patients considering total knee arthroplasty with preference report for surgeons: a pilot randomized controlled trial. BMC Musculoskelet Disord. 2014 Feb 24;15:54. doi: 10.1186/1471-2474-15-54. PMID 24564877
- [Background] Sepucha KR, Stacey D, Clay CF, Chang Y, Cosenza C, Dervin G, Dorrwachter J, Feibelmann S, Katz JN, Kearing SA, Malchau H, Taljaard M, Tomek I, Tugwell P, Levin CA. Decision quality instrument for treatment of hip and knee osteoarthritis: a psychometric evaluation. BMC Musculoskelet Disord. 2011 Jul 5;12:149. doi: 10.1186/1471-2474-12-149. PMID 21729315
- [Result] Stacey D, Taljaard M, Dervin G, Tugwell P, O'Connor AM, Pomey MP, Boland L, Beach S, Meltzer D, Hawker G. Impact of patient decision aids on appropriate and timely access to hip or knee arthroplasty for osteoarthritis: a randomized controlled trial. Osteoarthritis Cartilage. 2016 Jan;24(1):99-107. doi: 10.1016/j.joca.2015.07.024. Epub 2015 Aug 4. PMID 26254238
- [Result] Trenaman L, Stacey D, Bryan S, Taljaard M, Hawker G, Dervin G, Tugwell P, Bansback N. Decision aids for patients considering total joint replacement: a cost-effectiveness analysis alongside a randomised controlled trial. Osteoarthritis Cartilage. 2017 Oct;25(10):1615-1622. doi: 10.1016/j.joca.2017.05.022. Epub 2017 Jun 15. PMID 28624294
- [Derived] Trenaman L, Stacey D, Bryan S, Payne K, Hawker G, Bansback N. Long-term effect of patient decision aids on use of joint replacement and health care costs. Osteoarthritis Cartilage. 2020 Jun;28(6):819-823. doi: 10.1016/j.joca.2020.01.019. Epub 2020 Mar 12. PMID 32173628